CLINICAL TRIAL: NCT06878729
Title: Antegrade Dissection and Re-entry Versus Retrograde Strategy in Chronic Total Occlusion Percutaneous Coronary Intervention
Brief Title: Antegrade Dissection and Re-entry Versus Retrograde Strategy in CTO PCI
Acronym: ADRENALINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/ABM/01/00006; 2024/ABM/01/00006 (Other: National Institute of Cardiology, Warsaw, Poland)
Record Dates: First submitted 2025-03-04; First posted 2025-03-17 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Coronary Occlusion; Percutaneous Coronary Intervention
Keywords: coronary artery disease; percutaneous coronary intervention; coronary chronic total occlusion; antegrade dissection and re-entry; retrograde strategy
MeSH Terms: conditions — Coronary Artery Disease; Coronary Occlusion

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either ADR or retrograde CTO crossing strategy in a 1:1 fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADR strategy (Other): Patients with either failed or unattempted primary antegrade wiring strategy will be evenly randomized (1:1 fashion) to either ADR or retrograde CTO crossing strategy. The ADR, as part of the antegrade approach, involves extraplaque crossing of the occluded coronary artery with subsequent reentry into the distal true lumen using dedicated reentry systems or knuckle wire techniques.
  Interventions: Procedure: CTO PCI using ADR strategy
- Retrograde strategy (Other): Patients with either failed or unattempted primary antegrade wiring strategy will be evenly randomized (1:1 fashion) to either ADR or retrograde CTO crossing strategy. The retrograde technique, planned as the comparator to the ADR strategy, relies on crossing the occluded coronary artery from the distal vessel (i.e. against the original direction of blood flow). Retrograde CTO crossing is attempted either with retrograde intraplaque wiring or more frequently using the retrograde dissection and reentry techniques.
  Interventions: Procedure: CTO PCI using retrograde strategy

INTERVENTIONS:
Procedure: CTO PCI using ADR strategy — CTO recanalization using ADR performed as primary or secondary CTO PCI strategy (i.e. in case of unattempted or failed antegrade wiring, respectively).
  Arms: ADR strategy
Procedure: CTO PCI using retrograde strategy — CTO recanalization using retrograde approach performed as primary or secondary CTO PCI strategy (i.e. in case of unattempted or failed antegrade wiring, respectively).
  Arms: Retrograde strategy

SUMMARY:
The ADRENALINE trial has been designed as a multi-center, prospective randomized study to compare the procedural and periprocedural outcomes of coronary chronic total occlusion (CTO) percutaneous coronary intervention (PCI) using antegrade dissection and re-entry (ADR) versus retrograde strategy. Beyond the patient-oriented outcomes, the influence of the studied CTO PCI strategies on the stress levels among interventional cardiologists will be explored.

The main questions it aims to answer are as follows:

* What is the difference between ADR versus retrograde strategy with regard to total procedure time, the rates of successful guidewire crossing and periprocedural complications as well as stress levels experienced by interventional cardiologists?
* Is retrograde approach associated with higher rates of myocardial injury/infarction based on cardiac troponin/cardiac magnetic resonance (CMR) as compared with ADR?

Participants will undergo pre- and postprocedural laboratory testing (cardiac troponin, CK-MB), CMR for late gadolinium enhancement and health status assessment. Subjects undergoing successful CTO PCI using antegrade wiring strategy will be included in the observational arm.

DETAILED DESCRIPTION:
The ADRENALINE trial is planned as a multicenter, prospective randomized research experiment in patients with clinical indication for PCI of CTO. The target population will comprise patients with at least difficult CTO (J-CTO score ≥2) and angiographic equipoise for either ADR or the retrograde CTO recanalization strategy as evaluated by 2 independent CTO PCI operators. The pre-procedural assessment will comprise cardiac magnetic resonance (CMR) for late gadolinium enhancement, laboratory testing (cardiac troponin, creatine kinase-MB) and health status assessed by the Seattle angina questionnaire (SAQ) and the Rose Dyspnea Scale. Subsequently patients with either failed or unattempted primary antegrade wiring strategy will be evenly randomized (1:1 fashion) to either ADR or the retrograde CTO crossing strategy (n=74), while subjects undergoing successful antegrade wiring will be included in the observational arm (n=47). After CTO PCI, the cardiac troponin and creatine kinase-MB will be measured at 12 hours intervals (at least up to 24 hours), while CMR with late gadolinium enhancement will be repeated within 5 days post-procedure (including the observational arm). The health status of the study participants (SAQ and the Rose Dyspnea Scale) will be re-assessed at 3-months post-CTO PCI. In addition, to investigate the effect of the studied CTO PCI strategies on the occupational hazard of interventional cardiologists, the physical and mental stress levels experienced by CTO operators will be continuously monitored during the procedure. The co-primary endpoint is defined as: 1) total procedure time and 2) successful guidewire crossing through CTO. The secondary endpoints include: time of successful guidewire crossing through CTO, final technical success of CTO PCI, radiation dose, contrast volume, equipment cost, procedural complications, rate of periprocedural myocardial injury, rate of new myocardial infarction on CMR, quality of life, target lesion failure (cardiac death, target vessel-related myocardial infarction, and clinically-driven target lesion revascularization) at 3 months follow-up, and stress indices experienced by physicians during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* clinical indication for CTO PCI as determined by the local heart team (presence of angina or equivalent symptoms and/or documented ischemia or viability)
* at least difficult native CTO lesion with J-CTO difficulty score ≥2 points on invasive angiography
* angiographic suitability for both ADR and the retrograde strategy as assessed by 2 independent hybrid CTO PCI operators
* informed consent for participation in the study

Exclusion Criteria:

* <18 years of age
* acute myocardial infarction
* cardiogenic shock
* severe valvular disease
* estimated life expectancy <1 year
* contraindication to PCI
* contrast allergy
* positive pregnancy test or breast-feeding
* native CTO lesion with easy or intermediate difficulty score on invasive angiography (J-CTO score <2 points)
* lack of angiographic equipoise between the ADR and the retrograde strategy as assessed by 2 independent hybrid CTO PCI operators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Total procedure time | procedural (1 day)
  Total procedure time in minutes.
Successful guidewire crossing through CTO | procedural (1 day)
  Rate of successful guidewire crossing through CTO.

SECONDARY OUTCOMES:
Technical success | procedural (1 day)
  Achievement of Thrombolysis In Myocardial Infarction grade 3 flow in all ≥2.5-mm distal branches with <30% residual stenosis.
Time of successful guidewire crossing | procedural (1 day)
  Time of successful guidewire crossing through CTO in minutes defined as the time from starting ADR or the retrograde approach to the time of successful CTO recanalization using any technique.
Fluoroscopy time | procedural (1 day)
  Fluoroscopy time in minutes.
Radiation dose | procedural (1 day)
  Total radiation dose in Gy and mGycm2.
Contrast volume | procedural (1 day)
  Total contrast volume in mL.
Cost of CTO PCI | procedural (1 day)
  Total cost of CTO PCI procedure in PLN.
Number and type of procedural complications | procedural (1 day)
  Total number and specification of procedural complications (death, non-fatal myocardial infarction, cardiac tamponade requiring pericardiocentesis, coronary perforation, stroke, major bleeding according to Bleeding Academic Research Consortium).
Periprocedural myocardial injury | in-hospital (2-5 days)
  Any periprocedural myocardial injury based on the dynamics of cardiac troponin.
Periprocedural myocardial infarction | in-hospital (2-5 days)
  Any periprocedural myocardial infarction based on the dynamics of creatine kinase-MB/cardiac troponin and according to Fourth universal definition of myocardial infarction.
Myocardial infarction on CMR | in-hospital (2-5 days)
  Any new myocardial infarction as assessed on serial CMR with late gadolinium enhancement.
Target lesion failure | 3-months
  Total number of cardiac death, target vessel-related myocardial infarction or clinically-driven target lesion revascularization.
All-cause death | 3-months
  Any death observed.
Cardiac death | 3-months
  Any cardiac death observed.
Target vessel-related myocardial infarction | 3-months
  Any target vessel-related myocardial infarction observed.
Clinically-driven target lesion revascularization | 3-months
  Any clinically-driven target lesion revascularization observed.
CCS class | 3-months
  Quality of life assessed by the Canadian Cardiovascular Society (CCS) grading scale measuring the severity of exertional angina (it uses a scale from 1 to 4 where 1 means angina only occurs with strenuous, rapid or prolonged exertion, and 4 means angina is present at rest).
SAQ score | 3-months
  Quality of life assessed by the Seattle Angina Questionnaire comprising a 19-item questionnaire categorized into five scales (angina frequency, angina stability, physical limitations, treatment satisfaction, and disease-specific quality of life) with each scale transformed to a 0-100 score (the higher the score, the better the quality of life).
Dyspnea severity on the Rose Dyspnea Scale | 3-months
  Quality of life assessed by the Rose dyspnea scale questionnaire measuring dyspnea complaints or shortness of breath (it consists of a score from 0 to 4, where 0 means no dyspnea complaints and 4 means the patient has complaints during no or minimal physical effort).
Heart rate | operator-related (1 day)
  Mean heart rate of the first CTO operator throughout CTO PCI.
Mean arterial pressure | operator-related (1 day)
  Mean arterial pressure in mmHg of the first CTO operator throughout CTO PCI.
Systolic blood pressure | operator-related (1 day)
  Mean systolic blood pressure in mmHg of the first CTO operator throughout CTO PCI.
Diastolic blood pressure | operator-related (1 day)
  Mean diastolic blood pressure in mmHg of the first CTO operator throughout CTO PCI.
Blood glucose concentration | operator-related (1 day)
  Continuous blood glucose concentration monitoring in mmol/l of the first CTO operator throughout CTO PCI.
Brain activity monitoring | operator-related (1 day)
  Continuous brain activity monitoring via quantitative near infrared spectroscopy system assessing changes in relative concentrations of oxygenated and deoxygenated hemoglobin of the frontal cortex of the first CTO operator throughout CTO PCI.
Salivary cortisol concentration | operator-related (1 day)
  Salivary cortisol concentration in ng/mL of the first CTO operator measured at 30-min intervals throughout CTO PCI.
High-sensitivity cardiac troponin concentration | operator-related (1 day)
  Changes in the blood concentration of the high-sensitivity cardiac troponin (ng/L) pre- and post-CTO PCI in the first CTO operator.
Perceived Stress Scale score | operator-related (1 day)
  Stress level assessment in the first CTO operator adapted to CTO procedure and based on the Perceived Stress Scale score containing 10 questions with a 5-point answer scale ranging from 0 ('never') to 4 ('very often') - the minimum score is 0 (indicating no stress) and the maximum score is 40 (indicating the highest level of stress).

CONTACTS AND LOCATIONS:
Overall Officials: Maksymilian Opolski, Principal Investigator — National Institute of Cardiology
Locations (3):
- Poland (3):
  - National Institute of Cardiology, Warsaw, Warsaw
  - 1st Military Clinical Hospital, Lublin
  - Hospital of the Ministry of the Interior and Administration, Lublin